CLINICAL TRIAL: NCT00823277
Title: Indicators for the Metabolic Syndrome as Well as the Influence of Different Gen-polymorphs on Weightloss and the Maintenance of Lower Weight Among Children in Treatment for Overweight
Brief Title: Metabolic Syndrome and Gen-polymorphs Influence on Weightloss Among Children in Treatment for Overweight
Status: Completed | Type: Observational
Sponsor: Holbaek Sygehus (Other)
Collaborators: University of Copenhagen (Other); Hagedorn Research Institute (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jens-Christian Holm, MD, Ph.D., Zealand University Hospital
Other Study IDs: 130109; SJ-98
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Childhood Obesity; NAFLD (Non-alcoholic Fatty Liver Disease); Hypertension; Hyperlipidemia; Insulin Sensitivity
MeSH Terms: conditions — Pediatric Obesity; Non-alcoholic Fatty Liver Disease; Hypertension; Hyperlipidemias; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples of Whoole Blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Overweight and obese Children (BMI SDS > 90th percentile according to Danish BMI sheets) 5-20 Years of age. Recruited from the Paediatric department, University Hospital Holbaek, Region Zealand, Denmark, University of Copenhagen
  Interventions: Other: Chronic care multidisciplinary intervention of childhood obesity

INTERVENTIONS:
Other: Chronic care multidisciplinary intervention of childhood obesity — Overweight and obese Children, 5-20 Years old, followed by Paediatricians and other Health Personals (multidisciplinary team). Included at their first visit in the clinic (baseline)and follow-up after ~ 1 Year.

SUMMARY:
Definition:

the overall objective is to examine childhood obesity with focus on NAFLD and its treatment. Further, we aimed to investigate the impact of genetic variation on obesity.

The specific aims are to;

* describe the degree of NAFLD among overweight and obese, Danish children. (hypothesis; the degree for pediatric NAFLD among Danish Children was equal that found in other Caucasian paediatric study populations).
* investigate the effect of a multidisciplinary intervention treatment of 1 year on liver fat content.

(hypothesis; the intervention could reduce the liver fat percentage and a reduction in BMI SDS would associate with a reduction in liver fat content) - Analyze changes in liver fat content in relation to changes in levels of fasting blood variables to see if any of them could be used as a clinical tool for monitoring hepatic steatosis in the clinic.

(hypothesis; serum aminotransferases (separately and their ratio, respectively), serum insulin, and HOMA-IR could predict improvement in liver fat content

- Investigate the association between genetic variants and obesity.

ELIGIBILITY:
Inclusion Criteria:

* 5- 20 Years old.
* Adipose. BMI > 90 % percentile
* New patient in the Children's Obesity Clinic, Paediatric Department, University Hospital Holbaek,Region Zealand, Denmark
* Informed Consent

Exclusion Criteria:

* Drop-outs

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Overweight and obese Children. 5-20 Years old. Paediatric Department, University Hospital Holbaek,Region Zealand, University of Copenhagen, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
weightloss | 1 Year

SECONDARY OUTCOMES:
NAFLD (non-alcoholic Fatty Liver Disease).Gene-polymorphs | 1 Year
  Nafld measured by Magnet resonance spectroscopy. Sequencing of MC4R

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe S. Bille, MD, Principal Investigator — Paediatric department, University Hospital Holbaek, Region Zealand, University of Copenhagen, Denmark
Locations (1):
- The Children's Obesity Clinic, Paediatric Department, University Hospital Holbaek, Region Zealand, University of Copenhagen, Holbæk, Denmark

REFERENCES:
- [Result] Chabanova E, Bille DS, Thisted E, Holm JC, Thomsen HS. MR spectroscopy of liver in overweight children and adolescents: investigation of (1)H T(2) relaxation times at 3T. Eur J Radiol. 2012 May;81(5):811-4. doi: 10.1016/j.ejrad.2011.02.017. Epub 2011 Mar 4. PMID 21377308
- [Result] Chabanova E, Bille DS, Thisted E, Holm JC, Thomsen HS. (1)H MRS assessment of hepatic steatosis in overweight children and adolescents: comparison between 3T and open 1T MR-systems. Abdom Imaging. 2013 Apr;38(2):315-9. doi: 10.1007/s00261-012-9930-2. PMID 22736224
- [Result] Bille DS, Chabanova E, Gamborg M, Fonvig CE, Nielsen TR, Thisted E, Thomsen HS, Holm JC. Liver fat content investigated by magnetic resonance spectroscopy in obese children and youths included in multidisciplinary treatment. Clin Obes. 2012 Feb;2(1-2):41-9. doi: 10.1111/j.1758-8111.2012.00038.x. Epub 2012 Apr 24. PMID 25586046